CLINICAL TRIAL: NCT01203371
Title: PHASE III, DOUBLE-BLIND, RANDOMIZED STUDY COMPARING THE EFFICACY AND SAFETY OF NAFTOPIDIL AND TAMSULOSIN TO TREATMENT THE SYMPTOMS OF LOWER URINARY TRACT IN PATIENTS WITH BENIGN PROSTATE HYPERPLASIA
Brief Title: Efficacy And Safety Study Of Naftopidil to Patients Treatment With LUTS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Apsen Farmaceutica S.A. (Industry)
Responsible Party: Apsen Farmacêutica S.A., Apsen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APS 001/2010; BRA10APS001
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hyperplasia
Keywords: naftopidil; symptoms of lower urinary tract; benign prostate hyperplasia; LUTS
MeSH Terms: conditions — Hyperplasia; Prostatic Hyperplasia | interventions — naftopidil; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naftopidil (Experimental): 0,25 mg (2 weeks) and 0,50 mg (10 weeks)
  Interventions: Drug: Naftopidil
- Tamsusolin (Active Comparator): 0,4 mg/day
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Naftopidil — 0,25 mg (2weeks) and 0,50 mg (10 weeks)
  Arms: Naftopidil
Drug: Tamsulosin — 0,4 mg/day
  Other Names: SECOTEX
  Arms: Tamsusolin

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of Naftopidil and Tamsulosin in the treatment of lower urinary tract symptoms through a comparative study of patients with benign prostatic hyperplasia.

DETAILED DESCRIPTION:
Inclusion Criteria:

Men ≥ 50 years Signs and symptoms of BPH A total IPSS of ≥ 10 Prostate volume of ≥20 mL (estimated by ultrasonography) PVR > 150mL

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 50 years
* Signs and symptoms of BPH
* IPSS of ≥ 10
* Prostate volume of ≥ 20 mL
* PVR > 150 mL

Exclusion Criteria:

* History of allergy to a AR antagonists
* Treatment with antiandrogen drugs
* Drugs with anticholinergic activity
* Significant history of orthostatic hypotension
* Concomitant neurological diseases
* Known or suspected neurogenic bladder dysfunction
* Carcinoma of the prostate or bladder
* Previous surgery for BPH or bladder neck obstruction
* History of recurrent UTI
* Concomitant active UTI

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2012-01-01 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score | 2, 4, 8 and 12 weeks

SECONDARY OUTCOMES:
Adverse Effect | 2, 4, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, Brazil